CLINICAL TRIAL: NCT04475250
Title: Train-of-four Monitoring Using the Tetragraph Neuromuscular Transmission Monitor and Comparison to Standard (Visual) Train-of-four Assessment With a Peripheral Nerve Stimulator
Brief Title: Train-of-four Monitoring Using the Tetragraph
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joseph D. Tobias (Other)
Responsible Party: Sponsor-Investigator, Joseph D. Tobias, Chairman, Dept. of Anesthesiology & Pain Medicine, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY00001075
Record Dates: First submitted 2020-07-13; First posted 2020-07-17 (Actual); Results first posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Tetragraph (Experimental)
  Interventions: Device: Tetragraph (TM) NMT Monitor

INTERVENTIONS:
Device: Tetragraph (TM) NMT Monitor — TetraGraph is a unique, EMG-based portable device for quantitative (objective) monitoring of neuromuscular function. It is a precise and easy to use tool for monitoring depth of block, ensuring adequate recovery of muscle function, and aiding the clinician to reduce the incidence of residual block.

SUMMARY:
This is a prospective study that will evaluate the feasibility of using the Tetragraph Neuromuscular Transmission Monitor in comparison to standard (visual) train-of-four assessment with a peripheral nerve stimulator in pediatric patients undergoing surgery.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients requiring anesthetic care and use of neuromuscular blockade
* Weight range of 20 - 60 kg

Exclusion Criteria:

* Patients with history of a peripheral neurologic or neuropathic disorder
* Patients in whom the upper extremity cannot be used for TOF monitoring
* Patients undergoing a surgical procedure in which neuromuscular blockade is not required
* Edematous patients

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-05-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tobias JD, Epstein RH, Rice-Weimer J, Yemele Kitio SA, Brull SJ, Kalsotra S. Pediatric Intraoperative Electromyographic Responses at the Adductor Pollicis and Flexor Hallucis Brevis Muscles: A Prospective, Comparative Analysis. Anesth Analg. 2024 Jul 1;139(1):36-43. doi: 10.1213/ANE.0000000000006926. Epub 2024 Jun 17. PMID 38885397

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tetragraph
Started | 100
Completed | 100
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Tetragraph
Number analyzed (Participants) | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 100
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 11 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 62
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 97
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 90
  More than one race | 4
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 100
Weight [Mean (Standard Deviation); unit: kilograms] | 39.5 (10.8)
Height [Mean (Standard Deviation); unit: centimeters] | 145 (16)
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 18.7 (3.3)

OUTCOME MEASURES:

1. Primary Outcome: Baseline TOFr (%)
Description: Train of four (TOF) is measured by giving 4 quick electrical pulses to the muscle and counting the number of muscle twitches. Baseline TOFr is the ratio between the fourth twitch of the train of four (TOF) sequence (T4) and the first (T1) prior to administration of the neuromuscular blocking agent and then multiplied by 100 to get a percentage. A lower TOFr equals stronger neuromuscular block and more muscle paralysis.
Time Frame: Immediately prior to start of surgery
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Tetragraph
Number analyzed (Participants) | 100
percent | 100.1 (8.4)

2. Primary Outcome: Recovered TOFr (%)
Description: Train of four (TOF) is measured by giving 4 quick electrical pulses to the muscle and counting the number of muscle twitches. Recovered TOFr is the ratio between the fourth twitch of the train of four (TOF) sequence (T4) and the first (T1) after recovery from the neuromuscular blocking agent and then multiplied by 100 to get a percentage. A TOFr greater than or equal to 90% indicates adequate recovery from the neuromuscular block.
Time Frame: At the end of surgery (maximum 7 hours from baseline)
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | Tetragraph
Number analyzed (Participants) | 100
percent | 90.1 (13.1)

3. Secondary Outcome: Baseline Amplitude (mV)
Description: The amplitude of the muscle action potential prior to administration of the neuromuscular blocking agent.
Time Frame: Immediately prior to start of surgery
Measure: Mean (Standard Deviation); unit: millivolts
Arm/Group | Tetragraph
Number analyzed (Participants) | 100
millivolts | 7.5 (2.4)

4. Secondary Outcome: Recovered Amplitude (mV)
Description: The amplitude of the muscle action potential after recovery from the neuromuscular blocking agent.
Time Frame: At the end of surgery (maximum 7 hours from baseline)
Measure: Mean (Standard Deviation); unit: millivolts
Arm/Group | Tetragraph
Number analyzed (Participants) | 100
millivolts | 6.5 (2)

5. Secondary Outcome: Rate of Muscle Recovery (Minutes)
Description: The amount of time it took to return to a TOFr >90% following reversal of neuromuscular blocking agent.
Time Frame: At the end of surgery (maximum 7 hours from baseline)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Tetragraph
Number analyzed (Participants) | 100
minutes | 2.6 (1.4)

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Tetragraph
All-Cause Mortality (participants affected / at risk) | 0/100
Serious Adverse Events (participants affected / at risk) | 0/100
Other Adverse Events (participants affected / at risk) | 0/100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-07): https://cdn.clinicaltrials.gov/large-docs/50/NCT04475250/Prot_SAP_000.pdf